CLINICAL TRIAL: NCT02457442
Title: Validation of the Interaction Model of the Anesthetic Potency of Sevoflurane, Propofol and Remifentanil
Brief Title: Interaction of Sevoflurane Propofol and Remifentanil in Anesthesia for Laparoscopic Surgery
Acronym: SPRV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SPRV; 157/15 (Other: KEK)
Record Dates: First submitted 2015-05-26; First posted 2015-05-29 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Drug Interactions; Anesthesia, Conduction
Keywords: Anesthetics, Inhalation; Anesthetics, Intravenous; Analgesics, Opioid
MeSH Terms: conditions — Respiratory Aspiration | interventions — Propofol; Remifentanil; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PR1 (Active Comparator): (Arm closed in May 2022) Propofol-Remifentanil: Prop high, Remi low. Changing Remi (up-and-down)
  Interventions: Drug: Propofol and Remifentanil
- PR2 (Active Comparator): (Arm closed in May 2022) Propofol-Remifentanil: Prop low, Remi high. Changing Prop (up-and-down)
  Interventions: Drug: Propofol and Remifentanil
- SR1 (Active Comparator): (Arm closed in May 2022) Sevoflurane-Remifentanil: Sevo high, Remi low. Changing Remi (up-and-down)
  Interventions: Drug: Sevoflurane and Remifentanil
- SR2 (Active Comparator): (Arm closed in May 2022) Sevoflurane-Remifentanil: Sevo low, Remi high. Changing Sevo (up-and-down)
  Interventions: Drug: Sevoflurane and Remifentanil
- SPR1 (Active Comparator): (Arm closed in October 2023) Sevoflurane-Propofol-Remifentanil: Sevo plus Remi intermediate, Remi intermediate; changing Propofol.
  Interventions: Drug: SPR 1
- SPR2 (Active Comparator): (Arm closed in October 2023) Sevoflurane-Propofol-Remifentanil: Sevo plus Remi intermediate, Remi intermediate; changing Sevoflurane.
  Interventions: Drug: SPR2

INTERVENTIONS:
Drug: Propofol and Remifentanil — High propofol and low remifentanil, changing remifentanil (up-and-down method)
  Arms: PR1
Drug: Propofol and Remifentanil — Low propofol and high remifentanil, changing propofol (up-and-down method)
  Arms: PR2
Drug: Sevoflurane and Remifentanil — High sevoflurane and low remifentanil, changing remifentanil (up-and-down method)
  Arms: SR1
Drug: Sevoflurane and Remifentanil — Low sevoflurane and high remifentanil, changing sevoflurane up-and-down method)
  Arms: SR2
Drug: SPR 1 — Triple combination with intermediate propofol and sevoflurane and intermediate remifentanil.
  SPR 1: Changing Propofol for skin incision.
  Arms: SPR1
Drug: SPR2 — Triple combination with intermediate propofol and sevoflurane and intermediate remifentanil.
  Changing Sevoflurane for skin incision.
  Arms: SPR2

SUMMARY:
Recently a new model for the interaction of sevoflurane propofol and remifentanil was developed. The potency of any combination of the three drugs is defined as probability that a subject tolerates laryngoscopy without movement response. The model allows to compare the potency of intravenous and inhalation anesthetics. If the model is valid also for other stimuli than laryngoscopy and for other responses (e.g. blood pressure or heart rate increase upon stimulation). If the model is valid equipotent concentrations of sevoflurane and propofol the same remifentanil concentration would be sufficient to suppress hemodynamic response to a given stimulus. This will be investigated it the study.

DETAILED DESCRIPTION:
Background

In general anesthesia propofol or volatile anesthetic are usually combined with opioids and the synergy between hypnotics and opioids is used to reduce the dose of each component in order to minimize side effects and to allow a rapid recovery. Current pharmacodynamic interaction models allow to estimate the potency of combinations of propofol and opioids, volatile anesthetics and opioids or propofol and sevoflurane respectively. In these interaction models the potency of the drug combinations is expressed as probability that motor response to laryngoscopy is suppressed (= tolerance of laryngoscopy, PTOL). The potency of the hypnotic drugs is represented by the concentration preventing motor response to laryngoscopy in 50% of the population (Ce50 hypnotic). Conversely potency of the opioids is represented as concentration reducing the Ce50 of the hypnotics by 50%.

The data of the three previous studies on propofol-remifentanil, propofol-sevoflurane and sevoflurane-remifentanil interaction were pooled and reanalyzed. The result was a triple interaction model of sevoflurane, propofol and remifentanil where sevoflurane and propofol were additive and either propofol or sevoflurane were synergistic with remifentanil. In contrast to the previous studies the response surface of the propofol-remifentanil and sevoflurane-remifentanil derived from the pooled re-analysis had a similar shape, which is reflected by a common C50 remifentanil and a common slope parameter. This means that remifentanil is equally synergistic to propofol and sevoflurane. The next step is to validate this interaction model with other stimuli than laryngoscopy and with other responses to stimulation that movement.

In clinical practice not motor response but hemodynamic response (heart rate and arterial blood pressure increase) upon surgical stimulation is used to titrate anesthetics and opioids.

In laparoscopic surgery after a small skin incision, carbon dioxide is inflated into the abdominal cavity to maintain an intraabdominal pressure of 14 mmHg. Recently the sevoflurane concentration preventing a heart rate or blood pressure increase greater than 20% upon installation of pneumoperitoneum (MAC BAR pneumoperitoneum) has been determined: The MAC BAR pneumoperitoneum (95% CI) of sevoflurane was 4.6 (4.3-4.9) without opioids and 2.4 (2.2-2.6) and 1.7 (1.4-2.1) vol% with an effect site remifentanil concentration of 1 and 2 ng ml-1.These values all correspond to 90% probability to tolerate laryngoscopy (PTOL) according to our triple interaction model (Hannivoort, BJA 2016), which indirectly supports our model.

The main purpose of this randomized controlled study is to validate our sevoflurane-propofol-remifentanil interaction model using skin incision and carbon dioxide insufflation (pneumoperitoneum) as stimulus and blood pressure and heart rate response as endpoint.

Objective

To determine the C50 remifentanil preventing a 20% increase of heart rate or mean arterial pressure upon installation of pneumoperitoneum at equipotent concentrations of sevoflurane or propofol To determine the C50 of sevoflurane and propofol preventing a 20% increase of heart rate or mean arterial pressure upon installation of pneumoperitoneum at a standardized concentration of remifentanil

To determine the C50 of propofol or sevoflurane preventing a 20% increase of heart rate or mean arterial pressure upon installation of pneumoperitoneum at standardized concentrations of remifentanil plus sevoflurane or propofol respectively.

Methods

Patients will be randomly assigned to six groups with different propofol sevoflurane and remifentanil target concentrations for skin incision: Two groups with be given propofol-remifentanil, sevoflurane-remifentanil and sevoflurane-propofol-remifentanil respectively. The up-and-down method will be applied to determine the C50ies. During surgery primarily remifentanil and secondarily sevoflurane or propofol are titrated to maintain mean arterial pressure and bispectral index within predefined limits.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1 or 2
* Written informed consent

Exclusion Criteria

* Cardiovascular disease
* Pulmonary disease
* Liver disease
* CNS disease
* Alcohol or drug abuse
* Chronic intake of CNS active drugs
* Body mass index > 35
* Diabetes mellitus
* Hypersensitivity or allergy to one of the study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
20% heart rate or mean arterial pressure increase upon installation of pneumoperitoneum | 5 Minutes upon establishment of intraabdominal working pressure (12 mmHg)

SECONDARY OUTCOMES:
Mean (SD) Bloodpressure during surgery | Values recorded on computer HD every 10 sec during anesthesia, expected to be on average ca. 60 - 240 minutes
Mean (SD) Bispectral Index during surgery | Values recorded on computer HD every 10 sec. during anesthesia, expected to be on average ca. 60 - 240 minutes
Mean (SD) Remifentanil concentration during surgery | During surgery, expected to be on average ca. 60 - 240 minutes
Postoperative quality of recovery score | During hospital stay, expected to be on average ca. 3-5 days

CONTACTS AND LOCATIONS:
Overall Officials: Martin Luginbühl, PD Dr. med., Study Chair — Spital Tiefenau, Inselgruppe, Abteilung für Anästhesie und Intensivmedizin
Locations (1):
- Department of Anesthesiology and Pain Therapy, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Schumacher PM, Dossche J, Mortier EP, Luginbuehl M, Bouillon TW, Struys MM. Response surface modeling of the interaction between propofol and sevoflurane. Anesthesiology. 2009 Oct;111(4):790-804. doi: 10.1097/ALN.0b013e3181b799ef. PMID 19741484
- [Background] Heyse B, Proost JH, Schumacher PM, Bouillon TW, Vereecke HE, Eleveld DJ, Luginbuhl M, Struys MM. Sevoflurane remifentanil interaction: comparison of different response surface models. Anesthesiology. 2012 Feb;116(2):311-23. doi: 10.1097/ALN.0b013e318242a2ec. PMID 22222473
- [Background] Luginbuhl M, Schumacher PM, Vuilleumier P, Vereecke H, Heyse B, Bouillon TW, Struys MM. Noxious stimulation response index: a novel anesthetic state index based on hypnotic-opioid interaction. Anesthesiology. 2010 Apr;112(4):872-80. doi: 10.1097/ALN.0b013e3181d40368. PMID 20216387
- [Background] Bouillon TW, Bruhn J, Radulescu L, Andresen C, Shafer TJ, Cohane C, Shafer SL. Pharmacodynamic interaction between propofol and remifentanil regarding hypnosis, tolerance of laryngoscopy, bispectral index, and electroencephalographic approximate entropy. Anesthesiology. 2004 Jun;100(6):1353-72. doi: 10.1097/00000542-200406000-00006. PMID 15166553
- [Background] Hannivoort LN, Vereecke HE, Proost JH, Heyse BE, Eleveld DJ, Bouillon TW, Struys MM, Luginbuhl M. Probability to tolerate laryngoscopy and noxious stimulation response index as general indicators of the anaesthetic potency of sevoflurane, propofol, and remifentanil. Br J Anaesth. 2016 May;116(5):624-31. doi: 10.1093/bja/aew060. PMID 27106965